CLINICAL TRIAL: NCT05555719
Title: Dentoskeletal Effects of Two Different Fixed Functional Appliances for Correction of Class II Malocclusion: A Comparative Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abo bakr fouad, Assistant lecturer, orthodontic department, Al Azhar university Cairo Boys, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 346/1137/16/10/19
Record Dates: First submitted 2022-09-21; First posted 2022-09-27 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Class II Malocclusion
Keywords: PowerScope; Mandibular Protraction Appliance
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: 2 treatment groups, both have class II malocclusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular Protraction Appliance (Experimental): the first group that received Mandibular Protraction Appliance
  Interventions: Device: Mandibular Protraction Appliance
- PowerScope Appliances (Experimental): the first group that received PowerScope Appliances
  Interventions: Device: PowerScope Appliance

INTERVENTIONS:
Device: Mandibular Protraction Appliance — Mandibular Protraction Appliance was installed on fixed orthodontic appliance
  Arms: Mandibular Protraction Appliance
Device: PowerScope Appliance — PowerScope Appliance was installed on fixed orthodontic appliance
  Arms: PowerScope Appliances

SUMMARY:
Fixed Functional Appliances comparisons in treatment of orthodontic class II malocclusion cases

DETAILED DESCRIPTION:
Comparison between two types of fixed functional appliances, the first one is the Mandibular Protraction Appliances, while the second one was the PowerScope Appliance.

the treatment duration was 6 months the patients age was considered according to Baccetti et al, CVMI 3,4

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal and dental class II malocclusion with mandibular retrognathia, SNB>= 4.
2. Patients in cervical vertebral maturation index 3 -5.
3. Age ranged from 13-16 years.
4. Overjet ≥ 5 mm.
5. Minimum crowding in dental arches requiring no extraction of any permanent teeth (excluding third molars).
6. Good oral hygiene and general health.
7. No previous orthodontic treatment or jaw's surgery.

Exclusion Criteria:

* Class I skeletal malocclusion
* periodontally compromised patient
* patients have systemic diseases interfering with orthodontic treatment

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
SNA angle (on Cephalometric radiograph) | 6 months
  Anteroposterior postition of maxilla in relation to the anterior cranial base (SN line)
SNB angle (on Cephalometric radiograph) | 6 months
  Anteroposterior postition of mandible in relation to the anterior cranial base (SN line)
ANB angle (on Cephalometric radiograph) | 6 months
  The relationaship between maxilla and mandible
Effective mandibular length (mm) (on Cephalometric radiograph) | 6 months
  the length of the mandible (change in length before and after treatment)
Mandibular plane angle (on Cephalometric radiograph) | 6 months
  the angle between inferior border of the mandible (Go Me) and the anterior cranial base (SN line)
Maxillary incisors inclination (angle) (on Cephalometric radiograph) | 6 months
  The change of maxillary incisors inclination between the long axis of most protruded upper incisors and anterior cranial base (Sn line)
Mandibular incisors inclination (angle) (on Cephalometric radiograph) | 6 months
  The change of mandibular incisors inclination between the long axis of most protruded upper incisors and anterior cranial base (Sn line)

SECONDARY OUTCOMES:
Upper lip retrusion (mm) (on Cephalometric radiograph) | 6 months
  the amount of upper lip retrusion in millimeter in relation to E line (line extended between pronasale and soft tissue pogonion points)
Lower lip protrusion (on Cephalometric radiograph) | 6 months
  the amount of lower lip protrusion in millimeter in relation to E line (line extended between pronasale and soft tissue pogonion points)

CONTACTS AND LOCATIONS:
Overall Officials: Abubakr M Fouad, Principal Investigator — Al-azhar university, Cairo - Egypt
Locations (1):
- Abubakr Mohamed Fouad, Cairo, Egypt